CLINICAL TRIAL: NCT06136741
Title: A Phase 2b, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Rezpegaldesleukin in the Treatment of Adult Patients With Moderate-to-Severe Atopic Dermatitis (REZOLVE-AD)
Brief Title: A Phase 2b Study to Evaluate Rezpegaldesleukin (Rezpeg) in the Treatment of Adult Patients With Moderate-to-Severe Atopic Dermatitis
Acronym: REZOLVE-AD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-358-05
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Moderate to Severe Atopic Dermatitis
MeSH Terms: interventions — rhoA GTP-Binding Protein

STUDY DESIGN:
Intervention Model Description: Patients will be randomized initially to 1 of 4 groups (A dose regimen, B dose regimen, C dose regimen, or D dose regimen [placebo]) for the blinded induction period. At Week 16, the start of the blinded maintenance period, patients who responded well to treatment will be re-randomized within their previously assigned groups to either maintenance regimen 1 or maintenance regimen 2. At Week 16, patients without an adequate response during the blinded induction period may be assigned to receive open label escape therapy through the maintenance period of the study (up to Week 52); however, patients receiving escape therapy with inadequate improvement in disease severity will be discontinued from the study therapy at Week 32. Any patients enrolled into the blinded maintenance period with acute exacerbation of atopic dermatitis may be eligible to receive open label escape therapy instead.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Arm A (Experimental): Rezpegaldesleukin Dose Regimen A every 2 weeks during the induction period
  Interventions: Drug: Rezpegaldesleukin
- Arm A1 (Experimental): Rezpegaldesleukin Dose Regimen A every 4 weeks during the maintenance period
  Interventions: Drug: Rezpegaldesleukin
- Arm A2 (Experimental): Rezpegaldesleukin Dose Regimen A every 12 weeks during the maintenance period
  Interventions: Drug: Rezpegaldesleukin; Drug: Placebo
- Arm B (Experimental): Rezpegaldesleukin Dose Regimen B every 4 weeks during the induction period
  Interventions: Drug: Rezpegaldesleukin; Drug: Placebo
- Arm B1 (Experimental): Rezpegaldesleukin Dose Regimen B every 4 weeks during the maintenance period
  Interventions: Drug: Rezpegaldesleukin
- Arm B2 (Experimental): Rezpegaldesleukin Dose Regimen B every 12 weeks during the maintenance period
  Interventions: Drug: Rezpegaldesleukin; Drug: Placebo
- Arm C (Experimental): Rezpegaldesleukin Dose Regimen C every 2 weeks during the induction period
  Interventions: Drug: Rezpegaldesleukin
- Arm C1 (Experimental): Rezpegaldesleukin Dose Regimen C every 4 weeks during the maintenance period
  Interventions: Drug: Rezpegaldesleukin
- Arm C2 (Experimental): Rezpegaldesleukin Dose Regimen C every 12 weeks during the maintenance period
  Interventions: Drug: Rezpegaldesleukin; Drug: Placebo
- Arm D (Placebo Comparator): Placebo every 2 weeks during the induction period
  Interventions: Drug: Placebo
- Arm D1 (Placebo Comparator): Placebo every 4 weeks during the maintenance period
  Interventions: Drug: Placebo
- Escape Therapy (open-label) (Experimental): Rezpegaldesleukin Dose Regimen A every 2 weeks during the maintenance period
  Interventions: Drug: Rezpegaldesleukin

INTERVENTIONS:
Drug: Rezpegaldesleukin — Pharmaceutical form: Injection solution Route of administration: subcutaneous
  Other Names: NKTR-358; REZPEG; LY3471851 (formerly)
  Arms: Arm A; Arm A1; Arm A2; Arm B; Arm B1; Arm B2; Arm C; Arm C1; Arm C2; Escape Therapy (open-label)
Drug: Placebo — Pharmaceutical form: Injection solution Route of administration: subcutaneous
  Arms: Arm A2; Arm B; Arm B2; Arm C2; Arm D; Arm D1

SUMMARY:
This is an interventional, randomized, parallel group, treatment, Phase IIb, double blind, 4-arm study to assess the effect of pegylated-recombinant-human interleukin-2 (rezpegaldesleukin) in adult participants with moderate to severe atopic dermatitis.

The estimated duration is 15-35 days for screening, an Induction Period of 16 weeks, a Maintenance Period from Week 16-Week 52, and a Posttreatment Follow-Up Period for an additional year up to approximately Week 104 for all patients. Patients with a response at Week 16 (end of induction therapy) will be re-randomized for the maintenance therapy period.

ELIGIBILITY:
Inclusion Criteria:

* Adults (from at least 18 years of age) with AD as defined by the American Academy of Dermatology Consensus Criteria for 1 year or longer prior to screening.
* AD disease severity at screening and randomization:

  * EASI of 16 or higher
  * IGA of 3 or 4
  * BSA of 10% or more
* Documented history, within 6 months prior to the screening visit, of either inadequate response or inadvisability of topical treatments.
* Able to complete patient questionnaires.
* Able and willing to comply with requested study visits and procedures.
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Prior use of systemic immune modulating therapies for AD (i.e., JAK inhibitors or biologics)
* Other skin conditions that would interfere with assessment of AD
* Treatment with a live (attenuated) immunization within 12 weeks prior to screening.
* Men and women (of reproductive potential) unwilling to use highly effective birth control and women who are pregnant or breastfeeding.
* Any malignancies or history of malignancies within 5 years prior to randomization (except for basal cell or squamous epithelial carcinomas of the skin that have been successfully treated with no evidence of metastatic disease for 3 years or cervical carcinoma in situ that has been successfully treated, with no evidence of recurrence within the 3 years prior to randomization).
* Known history of, or suspected, significant current immunosuppression, including history of invasive opportunistic infections despite infection resolution or otherwise recurrent infections of abnormal frequency or prolonged duration.
* Positive for human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) at screening.
* Severe concomitant illness that would in the Investigator's opinion inhibit the patient's participation in the study, including for example, but not limited to, hypertension, renal disease, neurological conditions, heart failure and pulmonary disease.
* Concurrent participation in any other investigational clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean percent change in the Eczema Area and Severity Index (EASI) from baseline at Week 16 | Week 0 and Week 16
  The EASI scores range from 0 to 72, with higher scores indicating more severe atopic dermatitis.

SECONDARY OUTCOMES:
Proportion of patients at week 16 achieving Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) of 0 or 1 and at least a 2-point reduction from their baseline value | Week 0 and Week 16
  The vIGA-AD scale ranges from 0 to 4, with higher score indicating more severe atopic dermatitis.
Proportion of patients at week 16 achieving a Eczema Area and Severity Index reduction of 75% relative to their baseline score (EASI-75) | Week 0 and Week 16
  The EASI scores range from 0 to 72, with higher score indicating more severe atopic dermatitis.
Proportion of patients at week 16 achieving a Eczema Area and Severity Index reduction of 90% relative to their baseline score (EASI-90) | Week 0 and Week 16
  The EASI scores range from 0 to 72, with higher score indicating more severe atopic dermatitis.
Proportion of patients at week 16 achieving a Eczema Area and Severity Index reduction of 50% relative to their baseline score (EASI-50) | Week 0 and Week 16
  The EASI scores range from 0 to 72, with higher score indicating more severe atopic dermatitis.
Proportion of patients at week 16 achieving a 4-point or greater improvement in Itch numerical rating scale (NRS) in the subset of patients with a 4-point or greater Itch NRS at baseline | Week 0 and Week 16
  The itch NRS goes from 0 to 10, with higher score indicating more severe itch.
Proportion of patients at week 16 achieving a SCORing Atopic Dermatitis Index (SCORAD) reduction of 75% from their baseline value | Week 0 and Week 16
  The SCORAD scores range from 0 to 103, with a higher score indicating more severe atopic dermatitis.
Proportion of patients at week 16 achieving a SCORAD reduction of 50% from their baseline value | Week 0 and Week 16
  The SCORAD scores range from 0 to 103, with a higher score indicating more severe atopic dermatitis.
Mean change from baseline over the period between week 0 and week 104 in Eczema Area and Severity Index (EASI) | From Week 0 through Week 104
  The EASI scores range from 0 to 72, with higher score indicating more severe atopic dermatitis.
Mean percent change from baseline over the period between week 0 and week 104 in Eczema Area and Severity Index (EASI) | From Week 0 through Week 104
  The EASI scores range from 0 to 72, with higher score indicating more severe atopic dermatitis.
Mean change from baseline over the period between week 0 and week 104 in SCORAD | From Week 0 through Week 104
  The SCORAD scores range from 0 to 103, with a higher score indicating more severe atopic dermatitis.
Mean percent change from baseline over the period between week 0 and week 104 in SCORAD | From Week 0 through Week 104
  The SCORAD scores range from 0 to 103, with a higher score indicating more severe atopic dermatitis.
Mean change from baseline over the period between week 0 and week 104 in body surface area (BSA) involvement | From Week 0 through Week 104
Mean percent change from baseline over the period between week 0 and week 104 in body surface area (BSA) involvement | From Week 0 through Week 104
Rezpegaldesleukin plasma concentration assessed throughout the study | Through end of study (week 104)
Incidence of Serious Adverse Events (SAEs) | Through end of study (week 104)
Incidence of Treatment Emergent Adverse Events (TEAEs) | Through end of study (week 104)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (87):
- United States (25):
  - Nektar Investigative Site, Bryant, Arkansas
  - Nektar Investigative Site, Fountain Valley, California
  - Nektar Investigative Site, Los Angeles, California
  - Nektar Investigative Site, Santa Monica, California
  - Nektar Investigative Site, Hialeah, Florida
  - Nektar Investigative Site, Hollywood, Florida
  - Nektar Investigative Site, Miami, Florida
  - Nektar Investigative Site, Miami Lakes, Florida
  - Nektar Investigative Site, St. Petersburg, Florida
  - Nektar Investigative Site, Tampa, Florida
  - Nektar Investigative Site, Marietta, Georgia
  - Nektar Investigative Site, Clarksville, Indiana
  - Nektar Investigative Site, Indianapolis, Indiana
  - Nektar Investigative Site, Louisville, Kentucky
  - Nektar Investigative Site, Flint, Michigan
  - Nektar Investigative Site, Troy, Michigan
  - Nektar Investigative Site, Las Vegas, Nevada
  - Nektar Investigative Site, New York, New York
  - Nektar Investigative Site, Fairborn, Ohio
  - Nektar Investigative Site, Mayfield Heights, Ohio
  - Nektar Investigative Site, Murfreesboro, Tennessee
  - Nektar Investigative Site, Bellaire, Texas
  - Nektar Investigative Site, Cypress, Texas
  - Nektar Investigative Site, Frisco, Texas
  - Nektar Investigative Site, Spokane, Washington
- Australia (7):
  - Nektar Investigative Site, Darlinghurst, New South Wales
  - Nektar Investigative Site, Kogarah, New South Wales
  - Nektar Investigative Site, Westmead, New South Wales
  - Nektar Investigative Site, Woolloongabba, Queensland
  - Nektar Investigative Site, Campbelltown, South Australia
  - Nektar Investigative Site, East Melbourne, Victoria
  - Nektar Investigative Site, Melbourne, Victoria
- Bulgaria (6):
  - Nektar Investigative Site, Sevlievo, Gabrovo
  - Nektar Investigative Site, Dupnitsa, Kyustendil
  - Nektar Investigative Site, Sofia, Sofia-Grad
  - Nektar Investigative Site, Lovech
  - Nektar Investigative Site, Pleven
  - Nektar Investigative Site, Sofia
- Canada (10):
  - Nektar Investigative Site, Calgary, Alberta
  - Nektar Investigative Site, Edmonton, Alberta
  - Nektar Investigative Site, Kelowna, British Columbia
  - Nektar Investigative Site, Surrey, British Columbia
  - Nektar Investigative Site, Barrie, Ontario
  - Nektar Investigative Site, Markham, Ontario
  - Nektar Investigative Site, Peterborough, Ontario
  - Nektar Investigative Site, Richmond Hill, Ontario
  - Nektar Investigative Site, Toronto, Ontario
  - Nektar Investigative Site, Québec, Quebec
- Croatia (3):
  - Nektar Investigative Site 5701, Zagreb, City of Zagreb
  - Nektar Investigative Site 5703, Zagreb, City of Zagreb
  - Nektar Investigative Site, Ivanić-Grad
- Czechia (3):
  - Nektar Investigative Site, Brno
  - Nektar Investigative Site, Pardubice
  - Nektar Investigative Site, Prague
- Germany (11):
  - Nektar Investigative Site, Augsburg, Bavaria
  - Nektar Investigator Site, Augsburg, Bavaria
  - Nektar Investigative Site, Erlangen, Bavaria
  - Nektar Investigative Site, Bad Bentheim, Lower Saxony
  - Nektar Investigative Site, Mainz, Rhineland-Palatinate
  - Nektar Investigative Site, Leipzig, Saxony
  - Nektar Investigative Site, Berlin
  - Nektar Investigative Site, Darmstadt
  - Nektar Investigative Site, Frankfurt
  - Nektar Investigative Site, Lübeck
  - Nektar Investigator Site, München
- Nektar Investigative Site, Gyula, Bekes County, Hungary
- Poland (16):
  - Nektar Investigative Site, Wroclaw, Lower Silesian Voivodeship
  - Nektar Investigative Site, Warsaw, Masovian Voivodeship
  - Nektar Investigative Site, Rzeszów, Podkarpackie Voivodeship
  - Nektar Investigative Site, Gdansk, Pomeranian Voivodeship
  - Nektar Investigative Site, Gdynia, Pomeranian Voivodeship
  - Nektar Investigative Site, Częstochowa
  - Nektar Investigative Site, Iława
  - Nektar Investigative Site, Katowice
  - Nektar Investigator Site, Krakow
  - Nektar Investigative Site, Krakow
  - Nektar Investigative Site, Lodz
  - Nektar Investigative Site, Poznan
  - Nektar Investigative Site, Szczecin
  - Nektar Investigative Site, Tarnów
  - Nektar Investigative Site, Warsaw
  - Nektar Investigative Site, Wroclaw
- Spain (5):
  - Nektar Investigative Site, Alicante
  - Nektar Investigative Site, Córdoba
  - Nektar Investigative Site, Granada
  - Nektar Investigative Site, Seville
  - Nektar Investigative Site, Zaragoza

IPD SHARING:
Plan to Share IPD: No